CLINICAL TRIAL: NCT04960943
Title: Efficacy and Safety of Pyrotinib in Patients With HER2 Positive Refractory or Metastatic Gastrointestinal Tumors
Brief Title: Efficacy and Safety of Pyrotinib in HER2 Positive Gastrointestinal Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, MD,PhD, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-HER2-G
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-02

CONDITIONS: Gastrointestinal Tumor; Effect of Drug
Keywords: pyrotnib, HER2, Gastrointestinal Tumor, Phase II
MeSH Terms: conditions — Digestive System Neoplasms | interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib (Experimental): Pyrotinib with or without paclitaxel/trastuzumab treatment
  Interventions: Drug: Pyrotinib with or without trastuzumab

INTERVENTIONS:
Drug: Pyrotinib with or without trastuzumab — After enrollment, patients of all the three cohorts were given 400 mg/d oral pyrotinib continuously, every 21 days as a cycle; Cohort 1 and 2 : Patients with gastric cancer or esophageal adenocarcinoma were combined with paclitaxel 80 mg/m2, intravenously, once on the first and eighth day. Cohort 3: Patients with colorectal cancer were given trastuzumab at an initial load dose of 8 mg/kg followed by 6 mg/kg every 3 weeks.
  Other Names: pyrotinib with other drugs

SUMMARY:
Targeting human epidermal factor receptor 2 (HER2) therapy have shown the anti-tumor efficacy in patients with HER2-positive gastrointestinal tumors. Pyrotinib is an irreversible small-molecule receptor tyrosine kinase inhibitor targeting both epidermal growth factor receptor (EGFR) and HER2. This study is designed to evaluate the efficacy and safety of Pyrotinib in patients with HER2 positive gastrointestinal tumors.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of Pyrotinib in patients with HER2 positive gastrointestinal tumors. Three cohorts were designed for this trial. Cohort 1: patients with gastric cancer or esophageal adenocarcinoma receiving paclitaxel combined with pyrotinib for second-line therapy; Cohort 2: patients with gastric cancer or esophageal adenocarcinoma receiving pyrotinib monotherapy for third-line or posterior line therapy; Cohort 3: patients with colorectal cancer receiving pyrotinib combined with/without trastuzumab for third-line or posterior line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18
2. ECOG performance status of 0 to 1.
3. Life expectancy of more than 12 weeks.
4. At least one measurable lesion exists.(RECIST 1.1) Histologically or cytologic confirmed HER2 positive gastrointestinal tumors who failed prior therapies.
5. Required laboratory values including following parameters:

   ANC: ≥ 1.5 x 10^9/L, Platelet count: ≥ 80 x 10^9/L, Hemoglobin: ≥ 90 g/L, Total bilirubin: ≤ 1.5 x upper limit of normal, ULN, ALT and AST: ≤ 1.5 x ULN, BUN and creatine clearance rate: ≥ 50 mL/min LVEF: ≥ 50% QTcF: < 470 ms
6. Signed informed consent.

Exclusion Criteria:

1. Subjects with third space fluid that can not be controled by drainage or other methods.
2. Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption.
3. Less than 4 weeks from the last radiotherapy, chemotherapy, target therapy
4. Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry. Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
5. Receiving any other antitumor therapy.
6. Known history of hypersensitivity to pyrotinib or any of it components. Ongoing infection (determined by investigator).
7. History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
8. Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
9. Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
10. Known history of neurological or psychiatric disease, including epilepsy or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-09-09 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  evaluated in the 24th month since the treatment began

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  evaluated in the 24th month since the treatment began

OTHER OUTCOMES:
overall survival(OS) | 24 months
  evaluated in the 24th month since the treatment began
time to progression (TTP) | 24 months
  time to progression since the treatment began
duration of response (DoR) | 24 months
  the time of duration of response
disease control rate (DCR) | 24 months
  the proportion of patients who had a best response
Safety and Tolerability | 24 months
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Zhu, phD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang J, Xu M, Wang C, Huang D, Zhang Z, Chen Z, Zhu X, Li W. Dual HER2 Targeted Therapy With Pyrotinib and Trastuzumab in Refractory HER2 Positive Metastatic Colorectal Cancer: A Result From HER2-FUSCC-G Study. Clin Colorectal Cancer. 2022 Dec;21(4):347-353. doi: 10.1016/j.clcc.2022.07.003. Epub 2022 Jul 16. PMID 35941028